CLINICAL TRIAL: NCT07181811
Title: Assessing the Effects of Ongoing Ocrelizumab (OCR) Therapy on Fatigue and Cognition in Veterans With Multiple Sclerosis: Utilizing Cognitive Assessment Scales, and Patient-Reported Outcome Measures
Brief Title: Assessing the Effects of Ongoing Ocrelizumab (OCR) Therapy on Fatigue and Cognition in Veterans With Multiple Sclerosis
Acronym: ML45855
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anza Memon (U.S. Federal Agency)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Anza Memon, Staff Neurologist- John D. Dingell VAMC, John D. Dingell VA Medical Center
Organization: John D. Dingell VA Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1841354-3; ML45855 (Other: John D. Dingell VA Medical Center)
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Veterans; MS; Cognitive assessment; Ocrelizumab; OCR; Modified Fatigue Impact Scale (MFIS); Brief International Cognitive Assessment for MS (BICAMS); multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Patients who have been on Ocrelizumab for at least one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocrelizumab Arm (Experimental): This is a prospective, interventional study involving 30 subjects who have been diagnosed with multiple sclerosis and being treated with Ocrelizumab for at least one year.
  Interventions: Other: Multiple Sclerosis patients who have been on Ocrelizumab will undergo cognitive and fatigue assessments

INTERVENTIONS:
Other: Multiple Sclerosis patients who have been on Ocrelizumab will undergo cognitive and fatigue assessments — The cognitive and fatigue assessments administered in this study are not currently part of the standard clinical care for multiple sclerosis patients on Ocrelizumab. By prospectively assigning participants to undergo these additional assessments, this aspect of the study is considered investigational, and findings may contribute to clinical decision-making regarding the incorporation of cognitive and fatigue assessments into routine management of multiple sclerosis conditions.
  Other Names: Modified Fatigue Impact Scale (MFIS); Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS)

SUMMARY:
This study seeks to assess the effects of long-term ocrelizumab therapy on fatigue (extreme tiredness) as well as cognition (thinking and reasoning skills, such as memory, learning and attention), in veterans with multiple sclerosis. The evaluation will involve cognitive assessment scales (to assess memory, attention and learning abilities), clinical evaluations (to assess nerve function and ability to move), and patient-reported outcome measures (in which you will answer questions about your tiredness, sleep and how you function in daily life).

These assessments will occur at baseline (visit 1), 6 month (Visit-2) and 12 months (visit 3) to track changes over time.

DETAILED DESCRIPTION:
This is a prospective, interventional study involving 30 subjects who have been diagnosed with multiple sclerosis (MS) and being treated with ocrelizumab (OCR) for at least one year. This study will be performed at the John D. Dingell, VA Medical Center. All participants will require full informed consent prior to any study- related procedures. All aspects of the study and informed consent forms will be reviewed and approved by the institutional Review Board (IRB). MS patients who have been on OCR- for MS treatment, and enrolled in this study will undergo cognitive and fatigue assessments using the Brief International Cognitive Assessment for MS (BICAMS) and the Modified Fatigue Impact Scale (MFIS), respectively. Importantly, the cognitive and fatigue assessments administered in this study are not currently part of the standard clinical care for MS patients on OCR. By prospectively assigning participants to undergo these additional assessments, this aspect of the study is considered investigational, and findings may contribute to clinical decision-making regarding the incorporation of cognitive and fatigue assessments into routine MS management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, men and women.
* Confirmed diagnosis of Multiple Sclerosis (MS) (relapsing or progressive forms).
* Expanded Disability Status Scale score between 0 and 7.5.
* On continuous ocrelizumab therapy for at least 1 year.
* Women of childbearing potential: Must agree to remain abstinent or use acceptable contraceptive methods during the study and for 6 months after the. last ocrelizumab dose; must have a negative pregnancy test before enrollment.

Exclusion Criteria:

* Patients without a confirmed diagnosis of MS based on McDonald 2017 Criteria.
* Not on ocrelizumab therapy for at least 6 months prior to study start.
* Currently receiving other disease-modifying therapies for MS in addition to Ocrelizumab.
* Experienced an MS relapse or corticosteroid use within the last 30 months prior to enrollment.
* History of major psychiatric conditions (severe depression, schizophrenia, bipolar disorder) interfering with assessments.
* Significant cognitive impairment due to non-MS-related conditions (Traumatic brain injury, dementia, other neurodegenerative diseases).
* Other major neurological disorders (e.g., Parkinson's, epilepsy, stroke).
* History of alcohol or substance abuse within the past year.
* Uncontrolled comorbidities (severe cardiovascular disease, diabetes with complications, renal/liver failure).
* Uncorrected vision or hearing impairments interfering with cognitive testing.
* Unable to provide informed consent due to cognitive or legal reasons.
* Pregnant, lactating, or planning to become pregnant during the study period.
* Currently enrolled in other interventional clinical trials affecting cognitive or fatigue outcomes.
* Known presence of recurrent or chronic infections (Human Immunodeficiency Virus, syphilis, tuberculosis).
* History or presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, Human T-lymphotropic virus type 1).
* Active bacterial, viral, fungal, mycobacterial infection requiring recent hospitalization or IV antibiotics.
* History of cancer (except treated basal cell, in situ squamous cell, or resolved cervical carcinoma).
* History of or currently active primary or secondary immunodeficiency.
* Severe allergic or anaphylactic reactions to monoclonal antibodies.
* Systemic autoimmune disorders causing progressive neurological disease (e.g., lupus, Sjögren's).
* Concomitant diseases requiring chronic systemic corticosteroid or immunosuppressant use.
* Significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease.
* History of other neurologic disorders (e.g., progressive multifocal leukoencephalopathy, central nervous system/spinal tumors, hereditary spastic paraparesis, mitochondrial encephalomyopathy, lactic acidosis, and stroke-like episodes syndrome, neuromyelitis optica-spectrum disorder).
* Recent systemic corticosteroid therapy within 4 weeks prior to baseline.
* Prior MS treatments with cyclophosphamide, mitoxantrone, or bone marrow transplant.
* Receipt of live, attenuated, or inactivated/component vaccine within 6 weeks before enrollment.
* Laboratory abnormalities: Positive hepatitis B markers, elevated liver enzymes (AST/ALT ≥2x ULN), cytopenias, low IgG/IgM.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive performance | Baseline to 12 months.
  Global cognitive performance will be assessed using a composite z-score, derived from 3 standardized tests:
  1. CVLT (California Verbal Learning Test): Measures verbal learning and memory. Immediate Recall Max score= 80, Min = 0. Short and Long-Delay Recall: Max = 16 each, Min = 0. Recognition: Max = 16, Min = 0. Higher scores = better memory and learning ability. Lower scores = memory/learning impairment.
  2. BVMT-R (Brief Visuospatial Memory Test-Revised): Measures visuospatial learning/ memory; 6 abstract designs × 3 learning trials.
     Max total learning = 36, Min = 0. Delayed Recall: Max = 12, Min = 0. Recognition: Max = 6, Min = 0. Higher = better visuospatial memory. Lower = difficulty in visual memory.
  3. SDMT (Symbol Digit Modalities Test): Measures information processing speed, attention, working memory.
  Max = 110, Min = 0. Higher = better processing, Lower = slower processing Individual raw scores will be standardized, averaged, and compared between baseline and 12 months.
Change in fatigue impact (Modified Fatigue Impact Scale, MFIS) | Baseline to 12 months.
  Change in total score on the Modified Fatigue Impact Scale (MFIS; 21 items). Item responses range 0-4 and total score ranges 0-84, with higher scores indicating greater fatigue impact.
  The outcome is the difference between MFIS total at baseline and over a 12-month period; higher score = greater fatigue impact (worse) and lower score = less fatigue impact (better).

SECONDARY OUTCOMES:
Change in health-related quality of life (Multiple Sclerosis Quality of Life-54; MSQOL-54, physical and mental composite scores) | Baseline to 12 months
  Change in the MSQOL-54 physical health composite and mental health composite scores (each transformed 0-100, higher = better). Scores are computed per MSQOL-54 scoring manual by transforming subscale raw scores to 0-100 scales and averaging the relevant subscales to produce the two composite scores. The outcome is the difference between baseline and 12-month composite scores for each domain; positive values indicate improvement in health-related quality of life.
Change in patient-reported physical and mental health (Patient-Reported Outcomes Measurement Information System, 29-item profile; PROMIS-29) | Baseline to 12 months
  Change in PROMIS-29 domain T-scores (physical function, fatigue, anxiety, depression, sleep disturbance, social roles, pain interference) and pain intensity (0-10).
  PROMIS domain scores are reported as T-scores (mean=50, SD=10); higher scores indicate greater symptom burden for negative domains (fatigue, pain, etc.) and better health for positive domains (physical function, social roles). The outcome will report domain-specific changes from baseline to 12 months; directionality is indicated per domain.
  Higher = worse for negative domains (anxiety, depression, fatigue, pain interference, sleep disturbance, pain intensity).
  Higher = better for positive domains (physical function, social roles).

CONTACTS AND LOCATIONS:
Locations (1):
- John D. Dingell VA Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The primary reasons are participant confidentiality and institutional restrictions. Although data will be de-identified for analysis, there remains a risk of re-identification, especially in small and sensitive populations such as veterans. In addition, participants will not consent to broad data sharing outside the research team.